CLINICAL TRIAL: NCT00945633
Title: Dietary, Physiological, Genetic, and Behavioral Predictors of Health in a Young, Ethnically-Mixed Population
Acronym: InSight
Status: Active, not recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 27036
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: Obesity; unhealthy weight gain
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival repository
Oversight: Data Monitoring Committee: No

SUMMARY:
Dietary intervention and other strategies to prevent unhealthy weight gain and the development of obesity should be based on knowledge of dietary, physiological, genetic and behavioral determinants and their contributing interactions. Identifying these determinants is difficult because physiological susceptibility to specific dietary and behavioral factors implicated in unhealthy weight gain differs between populations and individuals within the populations. The research challenge is identifying specific determinants in a free-living, adult population.

Understanding the interaction between diet and the underlying susceptibility factors such as physiologic, genetic and epigenetic, and behavioral factors mandate an integrated approach.

This integrated approach should include understanding the interplay of physiological factors (genetics, epigenetics, taste preferences, susceptibility to energy excess, etc.) and behavioral factors (food cravings, restraint, disinhibition, physical activity) as each of these domains is a potential driving force in energy expenditure, food preference, dietary choices, and food intake.

Which of these factor(s) is most important? The investigators propose that by examining dietary, physiological, genetic, and behavioral factors in an integrated fashion we will gain insight into the obesity epidemic and identify the most important determinants of weight gain. As a secondary aim, the investigators will identify a single parsimonious collection of factors and develop strategies to mitigate the risks of developing obesity.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, clinical study using an epidemiological approach. The sample consists of 90 free-living participants aged 20-35 years. The participants will undergo a series of assessments in the domains of diet, physiological factors, and behavioral factors at baseline and every 12 months for 2 years.

OBJECTIVES

1. Identify dietary, physiological, genetic and behavioral determinants of unhealthy weight gain in healthy, young, ethnically-mixed men and women.
2. Identify relationships between genetic measures of taste perception and the determinants of unhealthy weight gain in the said population.
3. Identify relationships among the determinants of unhealthy weight gain that contribute to an individual's susceptibility to obesity.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be healthy men and women between the ages of 20-35, with BMI < 27.5 kg/m2, and fasting blood glucose < 126 mg/dl.

Exclusion Criteria:

* History of diabetes, history of obesity (BMI > 30).
* History of known inherited medical conditions that might influence future health status.
* Current or planned medication usage that might influence future health status.
* Prior serious injuries/surgeries that might influence future health status.
* Women who are pregnant or breastfeeding (once enrolled, pregnancy will not cause subjects to be terminated from the study).
* Women who are < 6 months postpartal, or women who have discontinued breastfeeding < 3 months prior to screening.
* History of cancer (including skin cancer) within 5 years.
* History or organ transplant.
* Previous diagnosis with HIV, Hepatitis B or C, or tuberculosis.
* Abuse of alcohol or illegal drugs.
* Abnormal EKG.
* Presence of pacemaker, defibrillator, or implanted metal.
* History of eating disorders and abnormal psychological scores for the screening measures described under Psychological Assessment Measures in the Appendix. This psychological screening will be conducted approximately two weeks prior to outpatient testing.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample includes 90 free-living participants aged 20-35 years.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-06; Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | Annually over 2 years
  Changes in body weight (kg) from baseline

SECONDARY OUTCOMES:
Changes in fat mass | Annually over 2 years
  Changes in fat mass (kg) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Peter Katzmarzyk, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harrington DM, Martin CK, Ravussin E, Katzmarzyk PT. Activity related energy expenditure, appetite and energy intake: potential implications for weight management. Appetite. 2013 Aug;67:1-7. doi: 10.1016/j.appet.2013.03.005. Epub 2013 Mar 22. PMID 23523668
- [Result] Tudor-Locke C, Martin CK, Brashear MM, Rood JC, Katzmarzyk PT, Johnson WD. Predicting doubly labeled water energy expenditure from ambulatory activity. Appl Physiol Nutr Metab. 2012 Dec;37(6):1091-100. doi: 10.1139/h2012-097. Epub 2012 Sep 11. PMID 22963352
- [Result] Edwards LM, Kemp GJ, Dwyer RM, Walls JT, Fuller H, Smith SR, Earnest CP. Integrating muscle cell biochemistry and whole-body physiology in humans:(31)P-MRS data from the InSight trial. Sci Rep. 2013;3:1182. doi: 10.1038/srep01182. Epub 2013 Jan 31. PMID 23378914
- [Result] Staiano AE, Marker AM, Martin CK, Katzmarzyk PT. Physical activity, mental health, and weight gain in a longitudinal observational cohort of nonobese young adults. Obesity (Silver Spring). 2016 Sep;24(9):1969-75. doi: 10.1002/oby.21567. Epub 2016 Jul 28. PMID 27465398
- [Result] Raja GK, Sarzynski MA, Katzmarzyk PT, Johnson WD, Tchoukalova Y, Smith SR, Bouchard C. Commonality versus specificity among adiposity traits in normal-weight and moderately overweight adults. Int J Obes (Lond). 2014 May;38(5):719-23. doi: 10.1038/ijo.2013.153. Epub 2013 Aug 16. PMID 23949614
- [Result] Staiano AE, Martin CK, Champagne CM, Rood JC, Katzmarzyk PT. Sedentary time, physical activity, and adiposity in a longitudinal cohort of nonobese young adults. Am J Clin Nutr. 2018 Nov 1;108(5):946-952. doi: 10.1093/ajcn/nqy191. PMID 30475973
- [Result] Katzmarzyk PT, Most J, Redman LM, Rood J, Ravussin E. Energy expenditure and substrate oxidation in White and African American young adults without obesity. Eur J Clin Nutr. 2018 Jun;72(6):920-922. doi: 10.1038/s41430-018-0202-2. Epub 2018 May 30. PMID 29849180
- [Derived] Fazzino TL, Dorling JL, Apolzan JW, Martin CK. Meal composition during an ad libitum buffet meal and longitudinal predictions of weight and percent body fat change: The role of hyper-palatable, energy dense, and ultra-processed foods. Appetite. 2021 Dec 1;167:105592. doi: 10.1016/j.appet.2021.105592. Epub 2021 Jul 8. PMID 34245802
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151